CLINICAL TRIAL: NCT02595931
Title: Phase I Clinical Trial of M6620 (VX-970, Berzosertib) in Combination With the Topoisomerase I Inhibitor Irinotecan in Patients With Advanced Solid Tumors
Brief Title: M6620 and Irinotecan Hydrochloride in Treating Patients With Solid Tumors That Are Metastatic or Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01915; NCI-2015-01915 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCC 15-164; UPCI 15-164; HCC#15-164; 9938 (Other: UPMC Hillman Cancer Center LAO); 9938 (Other: CTEP); UM1CA186689 (NIH); UM1CA186690 (NIH); UM1CA186704 (NIH); UM1CA186717 (NIH)
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Colorectal Carcinoma; Metastatic Lung Small Cell Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Pancreatic Carcinoma; Refractory Colorectal Carcinoma; Refractory Lung Small Cell Carcinoma; Refractory Malignant Solid Neoplasm; Refractory Pancreatic Carcinoma; Stage III Colorectal Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Unresectable Colorectal Carcinoma; Unresectable Lung Small Cell Carcinoma; Unresectable Malignant Solid Neoplasm; Unresectable Pancreatic Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Small Cell Lung Carcinoma; Neoplasm Metastasis; Pancreatic Neoplasms; Lung Neoplasms | interventions — berzosertib; Specimen Handling; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (irinotecan, M6620) (Experimental): Patients receive irinotecan hydrochloride IV over 90 minutes and M6620 IV over 60 minutes on days 1 and 15. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy and collection of blood samples throughout the study and undergo CT at screening, throughout the study, and during follow up.
  Interventions: Drug: Berzosertib; Procedure: Biopsy Specimen; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Irinotecan Hydrochloride

INTERVENTIONS:
Drug: Berzosertib — Given IV
  Other Names: 2-Pyrazinamine, 3-(3-(4-((Methylamino)methyl)phenyl)-5-isoxazolyl)-5-(4-((1-methylethyl)sulfonyl)phenyl)-; M 6620; M6620; VX 970; VX-970; VX970
Procedure: Biopsy Specimen — Undergo biopsy
  Other Names: Biopsy Sample
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; CPT11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U 101440E; U-101440E; U101440E

SUMMARY:
This phase I trial studies the side effects and best dose of M6620 and irinotecan hydrochloride in treating patients with solid tumors that have spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable). M6620 and irinotecan hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of M6620 (VX-970, berzosertib) in combination with irinotecan hydrochloride (irinotecan) in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To estimate the safety and tolerability of M6620 (VX-970, berzosertib) in combination with irinotecan.

II. To document anti-tumor activity. III. To determine the pharmacokinetic (PK) and pharmacodynamic (PD) parameters of M6620 (VX-970, berzosertib) and irinotecan.

EXPLORATORY OBJECTIVE:

I. To identify molecular subpopulations of patients with increased sensitivity to the irinotecan and M6620 (VX-970, berzosertib) combination.

OUTLINE: This is a dose-escalation study.

Patients receive irinotecan hydrochloride intravenously (IV) over 90 minutes and M6620 IV over 60 minutes on days 1 and 15. Treatment repeats every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy and collection of blood samples throughout the study and undergo CT at screening, throughout the study, and during follow up.

After completion of study treatment, patients are followed up for 30 days, then at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed metastatic or unresectable malignancy that is refractory to standard therapy or for which no standard therapy exists and where irinotecan is deemed a reasonable treatment option
* FOR PATIENTS ENROLLED IN THE EXPANSION COHORT: Patients must have known deficiencies in the deoxyribonucleic acid (DNA)-Damage Response (DDR), e.g. mutations in ATM, PALB2, BRCA1/2 or other deficiencies after discussion with the Study Chair (prioritized), or patients can be enrolled with the following tumor types regardless of known DDR deficiency: pancreatic cancer, colorectal cancer, and small cell lung cancer
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral CT scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* No limit on prior lines of therapy for metastatic disease; prior adjuvant or neoadjuvant chemotherapy does not count as a prior line of therapy as long as completion of the adjuvant or neoadjuvant therapy was more than 1 year prior to patient enrollment
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of M6620 (VX-970, berzosertib) in combination with irinotecan in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky >= 70%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN); if liver involvement, =< 5 x ULN
* Creatinine clearance >= 60 mL/min/1.73 m^2
* Patients must have archived tumor tissue from prior tumor biopsy or surgical resections available for submission that is sufficient to complete molecular profiling
* FOR PATIENTS ENROLLED IN THE EXPANSION COHORT: Willingness to undergo mandatory biopsies (day -13, approximately 18 to 22 hours post end of irinotecan infusion and day 2, approximately 18 to 22 hours post end of irinotecan infusion [= 17 to 21 hours post end of M6620 (VX-970, berzosertib)]); patients enrolled to this cohort should have tumors deemed easily accessible for biopsies with low likelihood of complication
* The effects of M6620 (VX-970, berzosertib) on the developing human fetus are unknown; for this reason and because DNA-damage response (DDR) inhibitors may have teratogenic potential, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of M6620 (VX-970, berzosertib) administration

  * For this reason and because DNA-damage response (DDR) inhibitors may have teratogenic potential, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 6 months after study completion
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or other systemic therapy or radiotherapy or patients who have not recovered from adverse events due to prior administered agents as follows:

  * Chemotherapy < 4 weeks prior to entering the study
  * Radiotherapy < 4 weeks prior to entering the study
  * Nitrosoureas/mitomycin C < 6 weeks prior to entering the study
  * Targeted therapy < 2 weeks (or 5 half-lives, whichever is longer) prior to entering the study
  * Those who have not recovered from clinically significant adverse events due to prior agents administered to grade =< 1 or baseline, with exception of alopecia and peripheral neuropathy, unless approved by the protocol chair
  * Immunotherapy < 4 weeks prior to entering the study
* Patients who are receiving any other investigational agents
* Patients with unstable brain metastases should be excluded; however, patients with known brain metastases may participate in this clinical trial if they are clinically stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are on a stable or decreasing dose of steroids for at least 14 days prior to trial treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M6620 (VX-970, berzosertib) or irinotecan
* M6620 (VX-970, berzosertib) is primarily metabolized by CYP3A4; irinotecan and its active metabolite, SN-38, are metabolized by CYP3A4 and UGT1A1, respectively; therefore, concomitant administration with strong inhibitors or inducers of CYP3A4 should be avoided; valproic acid is known to inhibit the process of glucuronidation and may potentially enhance the toxicity of irinotecan; medications that enhance glucuronidation (i.e. phenytoin, phenobarbital, carbamazepine, rifampin, etc.) may also enhance clearance of SN-38, which may possibly decrease efficacy; therefore, concomitant administration of these drugs should be avoided; because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, severe active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; patients with chronic viral hepatitis may participate in this clinical trial if they are clinically stable with acceptable liver function
* Pregnant women are excluded from this study because M6620 (VX-970, berzosertib) as a DNA-damage response (DDR) inhibitor may have the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M6620 (VX-970, berzosertib), breastfeeding should be discontinued if the mother is treated with M6620 (VX-970, berzosertib); these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients with well-controlled disease, as determined by CD4 count and viral load, who are on antiretroviral therapy that does not contain a strong inducer or inhibitor of CYP3A4 (e.g. regimens containing ritonavir, cobicistat, efavirenz or etravirine) are allowed on trial; HIV-positive patients on combination antiretroviral therapy with strong inducers or inhibitors of CYP3A4 are ineligible because of the potential for pharmacokinetic interactions with M6620 (VX-970, berzosertib); patients with poorly controlled HIV are not eligible due to the increased risk of lethal infections when treated with marrow-suppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 28 days
  Will be defined as the highest dose level at which =< 20% patients experience dose limiting toxicity. A logistic regression model will be used to determine the MTD using all patients.
Recommended phase 2 dose (RP2D) of ATR kinase inhibitor M6620 (VX-970, berzosertib) and irinotecan hydrochloride | Up to 28 days
  The RP2D will be determined based on MTD and the feasibility of the administration.

SECONDARY OUTCOMES:
Incidence of adverse events of M6620 (VX-970, berzosertib) and irinotecan hydrochloride | Up to 6 months after completion of study treatment
  Will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. A toxicity will be considered to be an adverse event that is possibly, probably or definitely related to treatment. The maximum grade of toxicity for each category of interest will be recorded for each patient, and the summary results will be tabulated by category, grade, and dose level. Serious (>= grade 3) toxicities will be described on a patient-by-patient basis and will include any relevant baseline data.
Overall response rate | Up to 6 months after completion of study treatment
  Will be evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1. Tabulated by disease diagnosis and by dose level. Will also report the 95% confidence limits on the response rates. Will also report the response rate and confidence limits at that dose level separately.
Incidence of stable disease | Up to 6 months after completion of study treatment
  Tabulated by disease diagnosis and by dose level. Will also report the response rate and confidence limits at that dose level separately.
Progression-free survival | Duration of time from start of treatment to time of progression or death, whichever occurs first, assessed up 6 months after completion of study treatment
  Estimated using the Kaplan-Meier method and the corresponding 95% confidence interval will be provided.
Pharmacokinetic parameters of M6620 (VX-970, berzosertib) in combination with irinotecan hydrochloride | Days -14 through -11, 1, 2, and 15 through 18 of cycle 1 (each cycle = 28 days)
  Within-subject comparison of day 15 and day -14 irinotecan hydrochloride and SN38 area under the curve (AUC) and half-life (t1/2) will be performed. Maximum concentration (Cmax), AUC, t1/2, clearance (CL), and volume in steady state (Vss) of VX-970 with single-agent historical data at comparable doses will be compared. Induction of gamma H2AX as a marker of ATR-dependent replication stress in peripheral blood mononuclear cells (PBMCs) and tumor will be characterized.
Pharmacodynamic parameters of M6620 (VX-970, berzosertib) in combination with irinotecan hydrochloride | Up to day 15 of cycle 1 (each cycle = 28 days)
  Within-subject comparison of day 15 and day -14 irinotecan hydrochloride and SN38 AUC and t1/2 will be performed. Cmax, AUC, t1/2, CL, and Vss of VX-970 with single-agent historical data at comparable doses will be compared. Induction of gamma H2AX as a marker of ATR-dependent replication stress in PBMCs and tumor will be characterized.

OTHER OUTCOMES:
Change in biomarker levels | Baseline to up 6 months after completion of study treatment
  Paired t tests will be used to compare biomarker levels before and after treatment. The Benjamini and Hochberg's procedure will be used to control the false discovery rate at 30%. A descriptive analysis of patient tumor genotype and response to therapy will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Liza C Villaruz, Principal Investigator — University of Pittsburgh Cancer Institute LAO
Locations (23):
- United States (23):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee